CLINICAL TRIAL: NCT05795114
Title: Prevention of Perinatal Depression in Birthing People With a History of Adverse Childhood Experiences: A Type 2 Effectiveness Implementation Trial
Brief Title: Perinatal Depression and Adverse Childhood Experiences: Prevention Trial
Acronym: PPD-ACE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Emily Miller, Associate Professor, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STU00217940
Record Dates: First submitted 2023-03-10; First posted 2023-04-03 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Perinatal Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced treatment as usual (No Intervention): Those randomized to enhanced treatment as usual will receive brief psychoeducation about perinatal depression and the associations between ACEs and perinatal depression. Information about the collaborative care program will be provided. Individuals will be followed with monthly self-reported screens for depression, without any prevention programming for perinatal depression. Those identified to have incident depression symptoms will receive recommendations for treatment within the collaborative care model.
- ROSE intervention (Experimental): Those randomized to the intervention will be offered 4 group-based prenatal sessions and one individual postpartum "booster" session guided by the Reach Out, Stand Strong, Essentials for New Mothers (ROSE) program embedded within the collaborative care model. Participants will be followed with monthly self-reported screens for depression, and those identified to have incident depression symptoms will receive treatment within the collaborative care model.
  Interventions: Behavioral: Reach Out, Stand Strong, Essentials for New Mothers (ROSE) Program

INTERVENTIONS:
Behavioral: Reach Out, Stand Strong, Essentials for New Mothers (ROSE) Program — A 5-part interpersonal therapy based intervention
  Arms: ROSE intervention

SUMMARY:
The goal of this clinical trial is to evaluate the impact of ROSE in individuals with adverse childhood experiences. The main question it aims to answer is, compared to enhanced treatment as usual, does the delivery of ROSE within a collaborative care model improve depressive symptom trajectories and prevent the development of perinatal depression.

Participants will be randomized to either enhanced treatment as usual or the ROSE intervention, delivered by a care manager within a perinatal collaborative care program. They will complete self-reported surveys of their depression symptoms every 4 weeks to inform their symptom trajectories. They will also complete clinical interviews to establish any incident diagnoses of a major depressive episode.

DETAILED DESCRIPTION:
The salience of early life experiences during the transition to parenthood underscores the risk of perinatal depression for those with childhood adversity. Mitigation of the adverse effects of childhood adversity via prevention of perinatal depression is an essential component of a reproductive justice-focused public health strategy. Whether and how the collaborative care model can be most effectively leveraged to prevent perinatal depression among pregnant people with a history of ACEs is unknown. To answer these questions, investigators propose a randomized clinical trial of trauma-informed interpersonal therapy modeled after the ROSE intervention and embedded within a perinatal collaborative care program utilizing a type 2 hybrid effectiveness-implementation design.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* At least one prenatal visit at Northwestern Medicine
* Less than 24 weeks gestation
* Non-anomalous pregnancy
* English- or Spanish- speaking
* ACE score ≥ 2
* Singleton gestation

Exclusion Criteria:

* Intent to delivery outside of Prentice Women's Hospital
* Active major depressive episode
* Active substance use disorder
* Participation in a study with a competing intervention or outcome

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Depression symptoms | Up to 6 months postpartum
  Depression symptom trajectories will be measured via Patient Health Questionnaire-9 (PHQ-9) screens administered
Perinatal depression | Up to 6 months postpartum
  Perinatal depression includes any categorical diagnosis of a major depressive episode, assessed using the Longitudinal Interval Follow-Up Examination measured by trained research personnel masked to the intervention

SECONDARY OUTCOMES:
Anxiety symptoms | Up to 6 months postpartum
  Anxiety symptom trajectories will be measured via Generalized Anxiety Disorder-7 (GAD-7) screens administered every 4 weeks from enrollment until 6 months postpartum.
Generalized anxiety disorder | Up to 6 months postpartum
  Generalized anxiety disorder includes any categorical diagnosis of generalized anxiety disorder, assessed using the Longitudinal Interval Follow-Up Examination measured by trained research personnel masked to the intervention in the 3rd trimester, at 3 months postpartum, and at 6 months postpartum.
Post-traumatic stress disorder | Up to 6 months postpartum
  Post-traumatic stress disorder includes any categorical diagnosis of a post-traumatic stress disorder, assessed using the Longitudinal Interval Follow-Up Examination measured by trained research personnel masked to the intervention in the 3rd trimester, at 3 months postpartum, and at 6 months postpartum.
Perceived stress symptoms | Up to 6 months postpartum
  Stress symptom trajectories will be measured via Perceived Stress Scale (PSS) screens administered every 4 weeks from enrollment until 6 months postpartum.
  Minimum value: 0
  Maximum value: 40
  Higher scores indicate a worse outcome
General self-efficacy | Up to 6 months postpartum
  Self-efficacy will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Self-Efficacy scale, administered in the 3rd trimester, at 3 months postpartum, and at 6 months postpartum.
  Minimum value: 10
  Maximum value: 50
  Higher scores indicate a better outcome
Parenting self-efficacy | Up to 6 months postpartum
  Parenting self-efficacy will be measured with the Parenting Sense of Competence scale administered in the 3rd trimester, at 3 months postpartum, and at 6 months postpartum.
  Minimum value: 17
  Maximum value: 102
  Higher scores indicate a better outcome
Breastfeeding self-efficacy scale | Up to 6 months postpartum
  Breastfeeding self-efficacy will be measured with the Breastfeeding Self-Efficacy scale administered in the 3rd trimester, at 3 months postpartum, and at 6 months postpartum. Included are individuals who are breastfeeding at each of the assessed time-points.
  Minimum value: 14
  Maximum value: 70
  Higher scores indicate a better outcome
Attachment in adult relationships | Up to 6 months postpartum
  Attachment in adult relationships will be measured with the Experiences in Close Relationships-Revised Questionnaire administered in the 3rd trimester, at 3 months postpartum, and at 6 months postpartum.
Emotional support | Up to 6 months postpartum
  Emotional support will be measured with the PROMIS Emotional Support-Short Form administered in the 3rd trimester, at 3 months postpartum, and at 6 months postpartum.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No